CLINICAL TRIAL: NCT02336022
Title: The Evaluation of a Noninvasive Respiratory Monitor in Pediatric Patients Undergoing General Anesthesia
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Viviane Nasr, Anesthesiology, Boston Children's Hospital
Other Study IDs: IRB-P00015003
Record Dates: First submitted 2014-12-15; First posted 2015-01-12 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Respiratory Complications
Keywords: general anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: Respiratory Motion Inc

SUMMARY:
Pediatric postoperative patients are at increased risk for post-operative respiratory complications such as hypoventilation. There is no objective measure of early respiratory parameters that would predict respiratory compromise after surgery efficiently in pediatric patients. Current respiratory assessment in non-intubated patients relies on oximetry data, impendence respiratory rate monitor and subjective clinical assessment. Pulse oximetry has been extremely helpful in recognizing oxygen desaturations but it is a late indicator of respiratory decline. New advances in technology and digital signal processing have led to the development of an improved impedance based Respiratory Volume Monitor (RVM). The RVM (ExSpiron™, Respiratory Motion, Inc.; Waltham, MA) has been shown to provide accurate real-time, continuous, non-invasive measurements of tidal volume (TV), minute ventilation (MV) and respiratory rate (RR) mostly in adult patients. The investigators' primary hypothesis is that the non-invasive, impedance-based RVM monitor will accurately reflect TV, RR and MV in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients between the ages of 1 year and 17 years
* ASA status of 1-3
* scheduled to undergo a procedure with general anesthesia at Boston Children's Hospital

Exclusion Criteria:

* Patients undergoing an emergency procedure or a
* patients undergoing a procedure where the study monitor will interfere with the surgical procedure site or standard of care
* preexisting respiratory disease
* muscular disease affecting the respiratory system

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients undergoing general anesthesia for surgical procedures at Boston Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Respiratory rate accurately measured by the ExSpiron monitor during controlled ventilation. | intraoperative
Tidal Volume accurately measured by the ExSpiron monitor during controlled ventilation. | intraoperative
Minute ventilation accurately measured by the ExSpiron monitor during controlled ventilation. | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Viviane Nasr, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States